CLINICAL TRIAL: NCT03015051
Title: Randomized Controlled Trial to Compare the Efficacy of High Flow Nasal Cannula Oxygen Therapy vs Low Flow Oxygen Therapy in Bronchiolitis
Brief Title: High Flow Nasal Cannula vs Low Flow Oxygen Therapy in Bronchiolitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruiting subjects who meet the inclusion/exclusion criteria
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Luca Ronfani, Head of Clinical Epidemiology and Public Health Research Unit, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: High flow RCT
Record Dates: First submitted 2016-11-24; First posted 2017-01-09 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; High flow nasal cannula; Oxygen therapy
MeSH Terms: conditions — Bronchiolitis | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High flow (Experimental): High flow (2 L/kg/min) nasal cannula oxygen therapy
  Interventions: Drug: Oxygen
- Low flow (Active Comparator): Low flow (max 3 L/min) oxygen therapy
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen

SUMMARY:
Bronchiolitis is the most common respiratory infection of the lower respiratory tract that affects 11-12% of infants in their first year of life. Approximately 1-2% of patients with bronchiolitis require hospital admission because of poor feeding and/or breathing difficulties. The standard treatment for bronchiolitis is represented by oxygen-therapy and hydration while neither steroids nor epinephrine nor bronchodilators are recommended. One of the techniques of administration of oxygen in bronchiolitis is represented by the high flow (HFNC) or by a system in which oxygen is delivered to 2L/kg through nasal cannulas. The HFNC provides humidification, heating and oxygen, ensuring a minimum positive pressure, reduces breathing load and allows for better nutrition. The main aim of therapy with high flows is to reduce the days of oxygen therapy and the cases of intubation. However, up to now, there have been few studies on the use of HFNC in Pediatric Emergency Units. The Cochrane review on this topic, updated in May 2013, included only one randomized controlled trial (RCT) on a pilot study of 19 subjects comparing HFNC with oxygen administered via "head box". The oxygen saturation was higher in children HFNC after 8 (00% versus 96%, p=0.04) and 12 hours (99% vs 96%, p=0.04) but similar in both groups at 24 hours. The authors concluded that the available evidence is insufficient to determine the effectiveness of HFNC.

The aim of this study is to evaluate in a large number of cases the effectiveness of treatment with high flow versus standard treatment, in children with bronchiolitis referred to a Pediatric Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bronchiolitis
* age >28 days and <6 months
* Oxygen saturation (SaO2) <92%
* respiratory rate >60 breaths/min
* dyspnea with respiratory distress assessment instrument (RDAI) score ≥8
* daily milk or food intake less than 2/3 than normally assumed

Exclusion Criteria:

* chronic diseases or syndromes
* respiratory diseases (i.e. bronchopulmonary dysplasia)
* heart diseases
* preterm birth (before 36 weeks of gestational age)

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Hours of oxygen therapy | up to 5 days

SECONDARY OUTCOMES:
Number of subject admitted in intensive care unit | up to 5 days
Number of patients needing intubation | up to 5 days
Days of parenteral hydration or nasogastric enteral feeding | up to 5 days
  Number of days
Adverse events | up to 15 days
  Number and type. Frequency of possible complication such as pneumothorax, pneumomediastinum or atelectasis will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Barbi, MD, Study Chair — IRCCS Burlo Garofolo, Trieste, Italy; Stefania Norbedo, MD, Study Director — IRCCS Burlo Garofolo, Trieste, Italy
Locations (15):
- Italy (15):
  - Ospedale Maggiore, Bologna, Emilia-Romagna
  - Ospedale Morgagni-Pierantoni, Forlì, Emilia-Romagna
  - Ospedale Ravenna AUSL Romagna, Ravenna, Emilia-Romagna
  - Ospedale Santa Maria degli Angeli, Pordenone, Friuli Venezia Giulia
  - Pediatric Emergency Department, IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia
  - Ospedale Pediatrico IRCCS Bambino Gesú, Rome, Lazio
  - Istituto G. Gaslini, Genoa, Liguria
  - Fondazione MBBM c/o Ospedale San Gerardo, Monza, Lombardy
  - Ospedale A. Cardarelli, Campobasso, Molise
  - Ospedale Infantile Regina Margherita, Turin, Piedmont
  - Ospedale Castelli, Verbania, Piedmont
  - Ospedale Giovanni Paolo II, Olbia, Sardinia
  - Ospedale Provinciale di Macerata, Macerata, The Marches
  - Ospedale Principe di Piemonte Area Vasta 2, Senigallia, The Marches
  - Azienda Ospedaliera di Padova, Padua, Veneto

IPD SHARING:
Plan to Share IPD: Undecided